CLINICAL TRIAL: NCT05562817
Title: The Epidemiology , Health and Economic Burden of Respiratory Syncytial Virus Amongst Hospitalized Children Under 5 Years of Age in Jordan: National Multi-center Cross-sectional Study
Brief Title: The Epidemiology , Health and Economic Burden of RSV Amongst Hospitalized Children Under 5 Years of Age in Jordan
Acronym: RSV-JO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MENA Center for Research & Development and Internship (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Munir Abu-Helalah, Chief Medical Officer, MENA Center for Research & Development and Internship
Other Study IDs: RSV-Jo.Burden2022
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Jordan; Epidemiology; Clinical burden; Economic burden
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Financial Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RSV has a global healthcare burden and vaccine in the main preventive measure. There are no recent published studies that have evaluated the burden of RSV infections in the Middle East in term of incidence at a national level, complication rates, mortality rates, hospitalizations, secondary infections, or the direct and indirect costs. Most studies have been limited to identifying genotypes or calculating the incidence in selected sites. In order to facilitate the introduction of an effective preventive measure for control of RSV infections, it is essential at a national and regional levels to assess the burden of disease, molecular epidemiology, and economic burden based on direct and indirect costs of RSV infections.

DETAILED DESCRIPTION:
A Multi-center cross-sectional study. A total of 4 study centers will be included distributed in central, Northern and southern regions of Jordan as follows; 1. Princess Rahma Hospital for Children, Irbid, 2. Zarqa Hospital serving center and east of Jordan 3. Jordan University Hospital, Amman 4.Al Karak Public Hospital, Al Karak.

Case definition: 46 Diagnosis of acute respiratory infection: Defined as "an illness presenting with one or more of the following symptoms for less than 7 days: Fever, cough, earache, nasal congestion, rhinorrhea, sore throat, vomiting after coughing, Crackles, and labored, rapid or shallow breathing".

Study population:

Children <5 years of age admitted to study sites with

1. At least one sign of acute infection (temperature ≥38 °C or <35.5 °C, abnormal white blood cell [WBC] count or abnormal differential) and
2. At least 1 of the following respiratory signs or symptoms for less than 7 days: tachypnea, cyanosis, cough, sputum production, pleuritic chest pain, hemoptysis, dyspnea, sore throat. cough, runny nose, grunting, wheeze, apnoea, difficulty in breathing.

The main sample of 1000 children will be from hospitalized children The focus on the hospitalized patients to assess the role of RSV infections in hospitalization, complications and economic burden.

An additional sample of 200 children from emergency department and a representative outpatients or healthcare center at sample from emergency and outpatients clinics at Princess Rahma Governmental Hospital in Irbid and Jordan University Hospital in Amman, to assess the proportion of RSV positivity and cost burden of the visit.

This will be conducted at sample from emergency and outpatients clinics at Princess Rahma Governmental Hospital in Irbid and Jordan University Hospital in Amman.

Sample collection and processing:

* Nasopharyngeal (NP) specimen will be collected from each patient, who meets inclusion criteria and consent for the study, using NP swab then Multiplex viral (RT)PCR will be performed on each Nasopharyngeal specimen testing
* PCR will be used to diagnosed cases with RSV at the included sites.
* RSV positive samples will be further analyzed for genotyping.

Packaging and shipment of clinical specimens Specimens for virus detection from nasopharyngeal and oropharyngeal will be collected using Dacron or polyester flocked swabs in a viral transport medium (VTM) containing antifungal and antibiotic supplements. Specimens will be transported to the laboratory as soon as possible after collection. Specimens that cannot be delivered promptly to the laboratory will be stored and shipped at 2-8°C for up to 3 days.. For the Bronchoalveolar lavage, the same as applied on the nasopharyngeal and oropharyngeal specimens except that the storage 2-8°C will be up to 2 days and at - 20°C or ideally -70°C and shipped on dry ice if further delays are expected for more than 2 days. 50,51

* Samples will be analyzed at central laboratory using the same kits throughout the study.
* Multiplex viral (RT)PCR will be performed on each Nasopharyngeal specimen testing for respiratory viruses, namely:

  4 Viruses + RSV genotyping
* Flu A
* Flu B
* RSV-A
* RSV-B
* SARS-CoV-2
* Quality assurance measures will be performed throughout the study.
* Pharmacoeconomics data:The economic burden of RSV will be assessed. Applying societal perspective, all direct medical, direct non-medical and indirect costs will be quantified (collected). With micro-costing approach, multiplication of utilization of resource quantity and unit cost will be used. At first, all required resources to treat an episode of RSV cases will be identified, through including the quantity and/or frequency of medications, medical supplies, diagnostic tests, number of hospital bed days, ambulatory clinic visits, travel time and cost, work absence (hours or days absent) and/or productivity losses of caregivers, and informal care visits.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria:

A.-Patients age less than 5 years permanently resident in the study areas - hospitalized with acute respiratory infection according to below definition and criteria: hildren <5 years of age admitted to study sites with

1. At least one sign of acute infection (temperature ≥38 °C or <35.5 °C, abnormal white blood cell [WBC] count or abnormal differential) and
2. At least 1 of the following respiratory signs or symptoms for less than 7 days: tachypnea, cyanosis, cough, sputum production, pleuritic chest pain, hemoptysis, dyspnea, sore throat. cough, runny nose, grunting, wheeze, apnoea, difficulty in breathing.

outpatients and emergency department is of value,

B-An additional sample of 200 children from emergency and outpatients clinics who meets above criteria.

Exclusion Criteria:

A. Not permanently resident in Jordan.

-

Ages: 0 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Case definition: Diagnosis of acute respiratory infection: Defined as "an illness presenting with one or more of the following symptoms for less than 7 days: Fever, cough, earache, nasal congestion, rhinorrhea, sore throat, vomiting after coughing, Crackles, and labored, rapid or shallow breathing".
  Study population:
  Children <5 years of age admitted to study sites with
  1. At least one sign of acute infection (temperature ≥38 °C or <35.5 °C, abnormal white blood cell [WBC] count or abnormal differential) and
  2. At least 1 of the following respiratory signs or symptoms for less than 7 days: tachypnea, cyanosis, cough, sputum production, pleuritic chest pain, hemoptysis, dyspnea, sore throat. cough, runny nose, grunting, wheeze, apnoea, difficulty in breathing.
  outpatients and emergency department is of value, An additional sample of 200 children from emergency department and outpatients who meet above criteria will be also enrolled.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
to measure epidemiological burden of RSV infection in Jordan among hospitalized children under 5 years of age, proportion of RSV infections along with showing the data for the age 0-24 months and 25-59 months | 9 months
  to measure the total epidemiological burden of RSV infection in Jordan among hospitalized children under 5 years of age, proportion of RSV infections along with showing the data for the age 0-24 months and 25-59 months separately.

SECONDARY OUTCOMES:
To measure the Odds ratio for risk factors of RSV infections | 9 months
  To measure the odds ratio for risk factors for RSV infection: (Infants: especially premature infants or babies who are 6 months or younger, congenital heart disease, chronic respiratory disease such as cystic fibrosis, immune deficiency: primary or secondary to medical condition or treatment), neuromuscular disorders, such as muscular dystrophy)
To measure selected clinical characteristics of RSV infections requiring hospital admissions and complications rates | 9 months
  To measure the rates of clinical characteristics of RSV infections requiring hospital admissions and complications rates: duration of hospitalization, reason for admission, hypoxia, ICU admissions, pneumonia, ventilation, respiratory failure, Otitis media perforate or not perforated, presence of secondary infections, readmission, mortality rate particularly amongst premature infants or immunocompromised patients.
To measure the proportion of RSV positivity amongst children hospitalized with acute respiratory infections. | 9 months
  To measure the proportion of RSV positivity amongst children hospitalized with acute respiratory infections.
To quantify the direct and indirect costs of RSV infections both at the community and hospital levels including readmissions, direct and indirect medical and societal costs: | 12 months
  To quantify the direct and indirect costs of RSV infections both at the community and hospital levels including readmissions, direct and indirect medical and societal costs:
To measure the distribution of RSV genotypes using representative national sample. | 6 months
  To measure the distribution of RSV genotypes using representative national sample.
To measure the positivity rate for RSV, without genotyping, amongst a selected sample from emergency and outpatients clinics | 9 months
  To measure the positivity rate for RSV, without genotyping, amongst a selected sample from emergency and outpatients clinics at Princess Rahma Governmental Hospital in Irbid and Jordan University Hospital in Amman to measure the health and cost burden. Follow up of these subjects for revisits or admissions will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Groothuis JR, Hoopes JM, Jessie VG. Prevention of serious respiratory syncytial virus-related illness. I: Disease pathogenesis and early attempts at prevention. Adv Ther. 2011 Feb;28(2):91-109. doi: 10.1007/s12325-010-0100-z. Epub 2011 Feb 4. PMID 21318606
- [Result] GBD 2016 Lower Respiratory Infections Collaborators. Estimates of the global, regional, and national morbidity, mortality, and aetiologies of lower respiratory infections in 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Infect Dis. 2018 Nov;18(11):1191-1210. doi: 10.1016/S1473-3099(18)30310-4. Epub 2018 Sep 19. PMID 30243584